CLINICAL TRIAL: NCT00000295
Title: Progesterone Treatment in Female Smokers
Brief Title: Progesterone Treatment in Female Smokers - 12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-12; P50-09259-12
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1999-04

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Progesterone

INTERVENTIONS:
Drug: Micronized Progesterone

SUMMARY:
The purpose of this study is to investigate progesterone effects in female smokers

DETAILED DESCRIPTION:
Limited research has been done on the effects of gender and menstrual cycle in response to drugs of abuse in humans. The main goal of this pilot study is to investigate the safety and tolerability of progesterone treatment in female nicotine users. In addition, plasma progesterone levels reached with a single 200 mg dose of progesterone treatment will be measured. The study will be a double-blind placebo controlled, crossover trial in which 12 female smokers who are in the early follicular phase of their menstrual cycle will be enrolled. Druing the experimental sessions, subjects will be given a single 200 mg dose of micronized progesterone or placebo and multiple blood samples will be obtained to measure the plasma levels of progesterone. Starting 2 hours after progesterone or placebo treatment, subjects will have a self-administration period that will last around 2.5 hours. We hypothesize that administration of 200 mg of progesterone will achieve plasma progesterone concentrations similar to those found in the luteal phase of the menstrual cycle, 3-30 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

Female subjects aged 21-45 years with a smoking history of at least 20 cigarettes daily for at least 1 year. In good health as verified by medical history, screening examination, and screening laboratory tests. Not pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods other than hormonal contraceptives.

Exclusion Criteria:

History of heart disease, peripheral vascular disease, COPD, liver diseases, abnormal vaginal bleeding, suspected or known breast malignancy, or any other medical condition which physician investigator deems inappropriate for subject participation. Use of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history. Amenorrhea. Current use of oral or other types of hormonal contraceptives. Abuse of alcohol or any other recreational or prescription drug. Regular use of any other tobacco products, including smokeless tobacco and nicotine products. Known allergy to progesterone or peanuts.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1999-04; Study Completion 2001-12

PRIMARY OUTCOMES:
Behavioral
Subjective
Biochemical

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States